CLINICAL TRIAL: NCT04303728
Title: Muscle Ultrasound as a Predictor of Functional Status in Spinal Cord Injury Patients
Brief Title: Use of Muscle Ultrasound to Predict Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DSRB 2019/00923
Record Dates: First submitted 2020-01-29; First posted 2020-03-11 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscle ultrasound (Experimental): Muscle ultrasound will be performed for the patient on admission and at 1-2 months from inpatient rehabilitation.
  Interventions: Diagnostic Test: Muscle ultrasound

INTERVENTIONS:
Diagnostic Test: Muscle ultrasound — The muscle thickness and muscle quality will be assessed on ultrasound

SUMMARY:
Establish if change from the baseline in ultrasound muscle parameters over 2 months of rehabilitation correlates with functional status of SCI patients at the end of rehabilitation

DETAILED DESCRIPTION:
Rehabilitation is the key to ambulatory recovery in patients with spinal cord injury, although only 25% of patients regain this ability despite current rehabilitation protocols. There is emerging evidence that intensive and prolonged rehabilitation, though costly and manpower intensive, may result in ambulatory recovery in patients previously thought to be non-ambulant. However, there are no suitable clinical biomarkers which can identify these group of patients who will benefit from this intervention.

Hence the aim is to establish if change from the baseline in ultrasound muscle parameters over rehabilitation correlates with functional status of SCI patients.

ELIGIBILITY:
Inclusion Criteria:

1. First ever acute SCI
2. Age 21-65 years
3. Presence of weakness in the lower limbs (defined as either ASIA A, B, C or D)
4. Independent in ambulation prior to onset of SCI
5. Able to understand study procedures and sign informed consent
6. Clinical suitability for rehabilitation

Exclusion Criteria:

1. Presence of premorbid lower musculoskeletal conditions eg contractures, fractures, previous operations, that prevents proper ultrasound assessment of the affected limb
2. Cardiorespiratory conditions eg congestive cardiac failure (EF<40%), chronic arrhythmias, COPD stage 3-4
3. End stage illness, end stage renal failure, life expectancy <6 months
4. Other active neurological conditions
5. Botulinum toxin injection over the past 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Functional Independence Score | Baseline (Performed on admission to inpatient rehabilitation)
  An 18-item of physical, psychological and social function (graded from 1-7)
Functional Independence Score | Performed at 1-2 months after starting rehabilitation
  An 18-item of physical, psychological and social function (graded from 1-7)
Functional Independence Score | Performed at 3-6 months
  An 18-item of physical, psychological and social function (graded from 1-7)
Functional Independence Score | Performed at 1 year
  An 18-item of physical, psychological and social function (graded from 1-7)
Spinal Cord Independence Measure (SCIM) III | Baseline (Performed on admission to inpatient rehabilitation)
  It is used by health care practitioners to assess and grade the functional status of a person based on the level of assistance he or she requires, in patients with spinal cord injury. Only the patient's indoor mobility subscore will be assessed from abilities, graded from 0-8.
Spinal Cord Independence Measure (SCIM) III | Performed at 1-2 months after starting rehabilitation
  It is used by health care practitioners to assess and grade the functional status of a person based on the level of assistance he or she requires, in patients with spinal cord injury. Only the patient's indoor mobility subscore will be assessed from abilities, graded from 0-8.
Spinal Cord Independence Measure (SCIM) III | Performed at 3-6 months
  It is used by health care practitioners to assess and grade the functional status of a person based on the level of assistance he or she requires, in patients with spinal cord injury. Only the patient's indoor mobility subscore will be assessed from abilities, graded from 0-8.
Spinal Cord Independence Measure (SCIM) III | Performed at 1 year
  It is used by health care practitioners to assess and grade the functional status of a person based on the level of assistance he or she requires, in patients with spinal cord injury. Only the patient's indoor mobility subscore will be assessed from abilities, graded from 0-8.
ASIA score | Baseline (Performed on admission to inpatient rehabilitation)
  This is an assessor administered test that systematically examines the dermatomes and myotomes in spinal cord patients through testing the strength and sensation
ASIA score | Performed at 1-2 months after starting rehabilitation
  This is an assessor administered test that systematically examines the dermatomes and myotomes in spinal cord patients through testing the strength and sensation
ASIA score | Performed at 3-6 months
  This is an assessor administered test that systematically examines the dermatomes and myotomes in spinal cord patients through testing the strength and sensation
ASIA score | Performed at 1 year
  This is an assessor administered test that systematically examines the dermatomes and myotomes in spinal cord patients through testing the strength and sensation
Walking Index for Spinal Cord Injury II (WISCI II) | Baseline (Performed on admission to inpatient rehabilitation)
  A walking scale used by health care practitioners to grade the walking ability of SCI patients.
Walking Index for Spinal Cord Injury II (WISCI II) | Performed at 1-2 months after starting rehabilitation
  A walking scale used by health care practitioners to grade the walking ability of SCI patients.
Walking Index for Spinal Cord Injury II (WISCI II) | Performed on 3-6 months
  A walking scale used by health care practitioners to grade the walking ability of SCI patients.
Walking Index for Spinal Cord Injury II (WISCI II) | Performed on 1 year
  A walking scale used by health care practitioners to grade the walking ability of SCI patients.

SECONDARY OUTCOMES:
Range of motion of elbow, hip and knee | Baseline (Performed on admission to inpatient rehabilitation)
  Range of motion of elbow, hip and knee
Range of motion of elbow, hip and knee | Performed at 1-2 months after starting rehabilitation
  Range of motion of elbow, hip and knee
Range of motion of elbow, hip and knee | Performed at 3-6 months
  Range of motion of elbow, hip and knee
Range of motion of elbow, hip and knee | Performed at 1 year
  Range of motion of elbow, hip and knee
Spasticity | Baseline (Performed on admission to inpatient rehabilitation)
  (2) Spasticity of the elbow flexors, knee extensors and ankle plantarflexors using the Modified Ashworth Scale, with a higher score indicating worse spasticity
Spasticity | Performed at 1-2 months after starting rehabilitation
  (2) Spasticity of the elbow flexors, knee extensors and ankle plantarflexors using the Modified Ashworth Scale, with a higher score indicating worse spasticity
Spasticity | Performed at 3-6 months
  (2) Spasticity of the elbow flexors, knee extensors and ankle plantarflexors using the Modified Ashworth Scale, with a higher score indicating worse spasticity
Spasticity | Performed at 1 year
  (2) Spasticity of the elbow flexors, knee extensors and ankle plantarflexors using the Modified Ashworth Scale, with a higher score indicating worse spasticity

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Tay, MD, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital Rehabilitation Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No